CLINICAL TRIAL: NCT03720847
Title: Ovarian Hormone Withdrawal and Suicide Risk: An Experimental Approach
Brief Title: Effect of Perimenstrual Ovarian Steroid Supplementation on Perimenstrual Suicidality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16-2078; K99MH109667 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-10

CONDITIONS: Suicidal Ideation
Keywords: Steroid hormones; Estradiol; Progesterone; Depression; Suicide
MeSH Terms: conditions — Suicidal Ideation; Depression; Suicide | interventions — Estradiol; Progesterone; Sugars

STUDY DESIGN:
Intervention Model Description: Crossover 2-Condition Placebo-Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identical placebos provided by the UNC investigational drug service.
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Active condition, then Inactive condition (Experimental): Beginning 7 days after ovulation, active treatment begins 7 days after ovulation with an estradiol transdermal patch (0.1 mg/24 hrs) applied to the skin weekly (spanning 14 days of treatment) along with (active) 100 mg oral micronized progesterone capsules taken twice daily by mouth for 14 days. A 1-month washout is observed. Then, beginning 7 days after ovulation, inactive placebo capsules will be taken twice daily by mouth along with the application of inactive clear patches applied to the skin weekly for 14 days.
  Interventions: Drug: Estradiol Transdermal Patch 0.1 mg/24 hrs; Drug: Oral Micronized Progesterone; Drug: Inactive Clear Patch; Drug: Placebo capsule
- Inactive condition, then active condition (Placebo Comparator): Beginning 7 days after ovulation, inactive placebo capsules will be taken twice daily by mouth along with the application of inactive clear patches applied to the skin weekly for 14 days. After completing a 1-month washout, active treatment begins 7 days after ovulation with an (active) estradiol transdermal patch applied to the skin weekly (spanning 14 days of treatment) along with (active) 100 mg oral micronized progesterone capsules taken twice daily by mouth for 14 days.
  Interventions: Drug: Estradiol Transdermal Patch 0.1 mg/24 hrs; Drug: Oral Micronized Progesterone; Drug: Inactive Clear Patch; Drug: Placebo capsule

INTERVENTIONS:
Drug: Estradiol Transdermal Patch 0.1 mg/24 hrs — Estradiol transdermal patch delivering 0.1 mg/24 hour administered by affixing to skin for 14 days starting on day 7 after ovulation
  Other Names: Climara
Drug: Oral Micronized Progesterone — 100 mg oral micronized progesterone taken orally twice daily for 14 days starting day 7 after ovulation
  Other Names: Prometrium
Drug: Inactive Clear Patch — Matching placebo patch administered by affixing to skin for 14 days starting on day 7 after ovulation
  Other Names: Placebo transdermal patch
Drug: Placebo capsule — Matching placebo capsules administered twice daily for 14 days starting day 7 after ovulation
  Other Names: Sugar pill

SUMMARY:
This within-person, crossover, 2-condition, placebo-controlled study compares the impact of two perimenstrual conditions on severity of suicidal symptoms in females with past-month suicidality but minimal risk of imminent suicide attempt. The two conditions are (1) natural perimenstrual withdrawal from estradiol and progesterone (during placebo), (2) perimenstrual stabilization of estradiol and progesterone using transdermal estradiol and oral micronized progesterone.

DETAILED DESCRIPTION:
A large number of observational studies have documented increased risk of suicide attempt, suicide death, and more lethal attempts during the perimenstrual (around menses) window of the female reproductive cycle; however, no experiments have investigated the causal role of ovarian steroid changes across the natural perimenstrual period in risk factors for acute suicidality. In response, the proposed experimental work investigates a causal role of perimenstrual withdrawal from the hormones estradiol (E2) and progesterone (P4) in previously-documented acute perimenstrual increases in suicidality.

Participants are 30 women between the ages of 18 and 45 with current suicidal ideation but minimal risk for suicide attempt. Using a placebo-controlled, crossover within-person design, the experiment tests the hypothesis that suicidality will be heightened during natural perimenstrual E2/P4 withdrawal (under placebo), but that experimental prevention of this perimenstrual E2/P4 withdrawal (with exogenous administration of E2/P4 hormones) will prevent these perimenstrual increases in suicidality and associated risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Ability to adhere to medication regimen
* Speaks English
* Assigned female at birth with intact ovaries
* Premenopausal
* Normal menstrual cycles between 25-35 days
* Under current care of an outpatient mental health provider with visits occurring at least once every 3 months.
* At least 1 year postpartum.
* Willing to use a barrier method of birth control during the study.
* Normal weight (BMI between 18-29)
* Must report at least some recent suicidal ideation (in the past month) at the time of recruitment.
* Must be categorized as having acceptably low imminent risk for suicidal crisis/attempt by a licensed clinical psychologist utilizing evidence-based clinical and research guidelines for imminent suicide risk management.

Exclusion Criteria:

* Must not be pregnant, breastfeeding, or trying to become pregnant.
* Must not be taking any form of exogenous hormones or hormonal intrauterine device, and must have ended previous use of hormonal preparations at least one month prior to the study.
* Must not have a personal history of any chronic medical condition, including but not limited to metabolic or autoimmune disease, epilepsy, endometriosis, cancer, diabetes, cardiovascular, gastrointestinal, hepatic, renal, or pulmonary disease, and no personal or first degree family history of thromboembolic events.
* Any current cigarette smoking is exclusionary.
* Must not report a history of clinical diagnosis or treatment for postpartum depression or premenstrual dysphoric disorder (Note: Premenstrual Dysphoric Disorder diagnosis must have been made based on prospective daily ratings).
* Must not report any history of manic episode, any history of psychotic symptoms, or current substance use disorder.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since the study is focused on the menstrual cycle, the study includes only those assigned female sex at birth.
Enrollment: 30 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tory A Eisenlohr-Moul, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Susan Girdler, PhD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC) at Chapel Hill.
Time Frame: 9 to 36 months following publication
Access Criteria: Following execution of a data use/sharing agreement with the University of North Carolina at Chapel Hill

REFERENCES:
- [Derived] Barone JC, Wenzel E, Alluri V, Moriarity D, Pinna G, Walsh E, Rubinow DR, Morrow AL, Eisenlohr-Moul TA. Effects of estrogen and progesterone on neuroactive steroids and cytokines in patients with suicidality. Psychoneuroendocrinology. 2023 Nov;157:106359. doi: 10.1016/j.psyneuen.2023.106359. Epub 2023 Aug 9. PMID 37611527
- [Derived] Owens SA, Schmalenberger KM, Bowers S, Rubinow DR, Prinstein MJ, Girdler SS, Eisenlohr-Moul TA. Cyclical exacerbation of suicidal ideation in female outpatients: Prospective evidence from daily ratings in a transdiagnostic sample. J Psychopathol Clin Sci. 2023 Aug;132(6):704-715. doi: 10.1037/abn0000838. Epub 2023 Jun 15. PMID 37326562
- [Derived] Eisenlohr-Moul TA, Bowers SM, Prinstein MJ, Schmalenberger KM, Walsh EC, Young SL, Rubinow DR, Girdler SS. Effects of acute estradiol and progesterone on perimenstrual exacerbation of suicidal ideation and related symptoms: a crossover randomized controlled trial. Transl Psychiatry. 2022 Dec 30;12(1):528. doi: 10.1038/s41398-022-02294-1. PMID 36585408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between November 15, 2016 and August 12, 2017. All participants were recruited via social media advertisements to participate in "a study on the biology of stress, depression, and suicidal thoughts". All participants were enrolled at the single site for the study: UNC Chapel Hill Psychiatry Department laboratories.
Period: Condition 1
Arm/Group | Active Condition, Then Inactive Condition | Inactive Condition, Then Active Condition
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout
Arm/Group | Active Condition, Then Inactive Condition | Inactive Condition, Then Active Condition
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 2
Period: Condition 2
Arm/Group | Active Condition, Then Inactive Condition | Inactive Condition, Then Active Condition
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants.
Arm/Group | Overall Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.56 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Perimenstrual Change in Self-Injurious Thoughts and Behaviors Interview (SITBI) Suicidal Ideation Score
Description: The SITBI is an interview designed to assess various aspects of suicidality, including ideation, planning, intent, and behavior. This outcome is a single item representing suicidal ideation severity from the SITBI interview which was measured as part of a daily questionnaire completed via smart phone. The question was: "Today, how intense were your thoughts of killing yourself?". Each day, individuals chose a response ranging from 0 (Not at All) to 4 (Severe). Values could range from 0 to 4, and higher values indicate more suicidal ideation. Perimenstrual change scores are calculated for each person in a given condition as the mean of scores in the perimenstrual phase (final seven days of medication use in that condition) minus the mean in the midluteal phase (7 days starting on the day of the positive ovulation test for that condition). Therefore, positive values represent a perimenstrual increase in symptoms, and negative values represent a perimenstrual decrease in symptoms.
Time Frame: Midluteal Baseline and Perimenstrual
Population: All participants who were exposed to either condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Estradiol + Progesterone: .1mg/day of transdermal estradiol + 100mg oral micronized progesterone twice daily (200mg/day).
- Placebos: placebo patch + placebo pills twice daily.
Arm/Group | Active Estradiol + Progesterone | Placebos
Number analyzed (Participants) | 28 | 29
units on a scale | -.05 (.44) | .35 (.18)
Statistical Analysis 1: Comparison: Active Estradiol + Progesterone vs Placebos; Test type: Superiority; p = .012, t-test, 2 sided; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Mean Difference (Final Values) = .26 — Positive estimated value indicates greater perimenstrual increase in symptoms in the placebo condition relative to the active condition

2. Primary Outcome: Perimenstrual Change in Self-Injurious Thoughts and Behaviors Interview (SITBI) Suicidal Planning Score
Description: The SITBI is an interview designed to assess various aspects of suicidality. This outcome is a single item representing suicidal planning from the SITBI interview was measured as part of a daily questionnaire via smart phone. The question was: "Today, how seriously did you consider acting on a suicide plan?". Each day, individuals chose a response from 0 (Not at All) to 4 (Severe). Values could range from 0 to 4, and higher values indicate more suicidal planning. Perimenstrual change scores are calculated for each person in a given condition as the mean of scores in the perimenstrual phase (final seven days of medication use in that condition) minus the mean in the midluteal phase (7 days starting on the day of the positive ovulation test for that condition). Therefore, positive values represent a perimenstrual increase in symptoms, and negative values represent a perimenstrual decrease.
Time Frame: Midluteal Baseline and Perimenstrual
Population: All participants who were exposed to either condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Estradiol and Progesterone: .1mg/day of transdermal estradiol + 100mg oral micronized progesterone twice daily (200mg/day).
Arm/Group | Active Estradiol and Progesterone | Placebos
Number analyzed (Participants) | 28 | 29
units on a scale | -.06 (.26) | .17 (.22)
Statistical Analysis 1: Comparison: Active Estradiol and Progesterone vs Placebos; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Test type: Superiority; p = .030, t-test, 2 sided; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Mean Difference (Final Values) = .21 — Positive estimated value indicates a greater perimenstrual increase in the outcome in the placebo condition relative to the active condition

3. Secondary Outcome: Perimenstrual Change in Beck Hopelessness Scale (BHS) Score
Description: Hopelessness is assessed with the Beck Hopelessness Scale, a 20-item self-report measure with true-false items that assess hopelessness and the extent of positive and negative beliefs about the future. This measure will be collected at the second lab visit in each condition (day 7 following ovulation). Summed scores range from 0 to 20. Scores provide a measure of the severity of self-reported hopelessness: 0-3 minimal, 4-8 mild, 9-14 moderate, and 15-20 severe. Higher values on the raw scale represent greater hopelessness. Perimenstrual change scores are calculated for each person in a given condition as the person's score at lab 2 (in the perimenstrual phase) minus the person's score at lab 1 (midluteal phase). Therefore, positive values represent degree of perimenstrual increase in symptoms, and negative values represent degree of perimenstrual decrease.
Time Frame: Day 7 of Each Condition (Lab 2)
Population: All participants who were exposed to either condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Estradiol and Progesterone | Placebos
Number analyzed (Participants) | 29 | 28
units on a scale | -.017 (2.42) | 1.37 (2.72)
Statistical Analysis 1: Comparison: Active Estradiol and Progesterone vs Placebos; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Test type: Superiority; p = .013, t-test, 2 sided; Mean Difference (Final Values) = 3.16 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Perimenstrual Change in Center for Epidemiological Studies Depression Scale (CES-D) Score
Description: The Center for Epidemiological Studies Depression scale (CES-D) includes 20 items that ask the person assessed to report his or her experience of mood symptoms. Instructions were modified such that symptoms were rated over the past week (rather than the standard 2 weeks). This measure will be collected at the second lab visit in each condition (day 7 following ovulation). Scores can range from zero to 60, with most persons attaining a score of 15 or less. Higher scores are considered worse. Perimenstrual change scores are calculated for each person in a given condition as the person's score at lab 2 (in the perimenstrual phase) minus the person's score at lab 1 (midluteal phase). Therefore, positive values represent degree of perimenstrual increase in symptoms, and negative values represent degree of perimenstrual decrease.
Time Frame: Day 7 of Each Condition (Lab 2)
Population: All participants who were exposed to either condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Estradiol and Progesterone | Placebos
Number analyzed (Participants) | 28 | 29
units on a scale | -1.53 (4.62) | 2.69 (7.89)
Statistical Analysis 1: Comparison: Active Estradiol and Progesterone vs Placebos; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Test type: Superiority; p = .018, t-test, 2 sided; Mean Difference (Final Values) = 3.65 — Positive estimated value indicates greater perimenstrual change in the placebo condition relative to the active condition

5. Secondary Outcome: Perimenstrual Change in Lack of Premeditation Subscale Score of the "Urgency, Premeditation, Perseverance, Sensation Seeking, and Positive Urgency (UPPSP) Impulsivity Scale"
Description: The UPPS-P (Urgency, Premeditation, Perseverance, Sensation Seeking, Positive Urgency Impulsivity Scale) Lack of Premeditation subscale includes 11 items that ask the person to report experience of impulsivity over the past two weeks. Instructions were modified such that symptoms were rated over the past week (rather than the standard 2 weeks). This measure will be collected at the second lab visit in each condition (day 7 following ovulation). Scores can range from 11 to 44. Higher scores are considered worse. Perimenstrual change scores are calculated for each person in a given condition as the person's score at lab 2 (in the perimenstrual phase) minus the person's score at lab 1 (midluteal phase). Therefore, positive values represent degree of perimenstrual increase in symptoms, and negative values represent degree of perimenstrual decrease.
Time Frame: Day 7 of Each Condition (Lab 2)
Population: All participants who were exposed to either condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Estradiol and Progesterone | Placebos
Number analyzed (Participants) | 29 | 28
units on a scale | -.75 (1.75) | .27 (2.43)
Statistical Analysis 1: Comparison: Active Estradiol and Progesterone vs Placebos; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Test type: Superiority; p = .073, t-test, 2 sided; Mean Difference (Final Values) = 1.04 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Perimenstrual Changes in Patient-Reported Outcomes Measurement Information Systems (PROMIS) Anxiety Scale Score
Description: The PROMIS (Patient-Reported Outcomes Measurement Information Systems) Anxiety scale includes 7 items that ask the person assessed to report his or her experience of anxiety over the past two weeks. Instructions were modified such that symptoms were rated over the past week (rather than the standard 2 weeks). This measure will be collected at the second lab visit in each condition (day 7 following ovulation). Scores can range from 7 to 35. Higher scores are considered worse. Perimenstrual change scores are calculated for each person in a given condition as the person's score at lab 2 (in the perimenstrual phase) minus the person's score at lab 1 (midluteal phase). Therefore, positive values represent degree of perimenstrual increase in symptoms, and negative values represent degree of perimenstrual decrease.
Time Frame: Day 7 of Each Condition (Lab 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Estradiol and Progesterone | Placebos
Number analyzed (Participants) | 28 | 29
units on a scale | 1.39 (2.80) | .17 (3.37)
Statistical Analysis 1: Comparison: Active Estradiol and Progesterone vs Placebos; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Test type: Superiority; p = .25, t-test, 2 sided; Mean Difference (Final Values) = -1.16

7. Secondary Outcome: Perimenstrual Change in State Self-Esteem Scale Social Evaluation Subscale (SSES-SE) Score
Description: The SSES-SE (State Self-Esteem Scale Social Evaluation subscale) includes 7 items that ask the person assessed to report his or her experience of social self-esteem--that is, a sense that others are evaluating one in a positive light-- in the present moment. Instructions were modified such that symptoms were rated over the past week (rather than the standard 2 weeks). This measure will be collected at the second lab visit in each condition (day 7 following ovulation). Scores can range from 7 to 49. Higher scores are considered better as they indicate better social self-esteem. Perimenstrual change scores are calculated for each person in a given condition as the person's score at lab 2 (in the perimenstrual phase) minus the person's score at lab 1 (midluteal phase). Therefore, positive values represent degree of perimenstrual increase in self-esteem, and negative values represent degree of perimenstrual decrease.
Time Frame: Day 7 of Each Condition (Lab 2)
Population: All participants who were exposed to either condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Estradiol and Progesterone | Placebos
Number analyzed (Participants) | 29 | 28
units on a scale | 1.65 (4.26) | -.33 (4.78)
Statistical Analysis 1: Comparison: Active Estradiol and Progesterone vs Placebos; paired sample t-test comparing perimenstrual change in the placebo vs. active conditions within a given participant; Test type: Superiority; p = .23, t-test, 2 sided; Mean Difference (Final Values) = -1.32

ADVERSE EVENTS:
Time Frame: The two weeks of patch/pill administration that occurred during each of the two conditions.
Description: Assessed during daily study phone calls. Under "Participant Flow", Arm/Group is represented by two condition order categories (i.e., "Active Condition, then Inactive Condition" vs. "Inactive Condition, then Active Condition"); this allows one to understand effects of condition order on participant flow. Here, Arm/Group is represented as exposure to active vs. placebo conditions, since that is the relevant grouping to understand how placebo vs. active medication influenced risk of adverse events.
Arm/Group | Active Estradiol + Progesterone | Placebos
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 15/28 | 18/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Estradiol + Progesterone (N=28) | Placebos (N=29)
Skin Itching (General disorders) | 8 (8) | 7 (7) — Itching around patch.
Breast Tenderness (General disorders) | 8 (8) | 8 (8)
Headache (General disorders) | 5 (5) | 9 (9)
Nausea (General disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT03720847/Prot_SAP_000.pdf